CLINICAL TRIAL: NCT03835780
Title: The Risk of Venous Thromboembolism in Systemic Inflammatory Disorders: a UK Matched Cohort Study
Brief Title: The Risk of Venous Thromboembolism in Systemic Inflammatory Disorders: a United Kingdom (UK) Matched Cohort Study
Status: Completed | Type: Observational
Sponsor: Momentum Data (Industry)
Collaborators: Pfizer (Industry); University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: P004
Record Dates: First submitted 2019-01-17; First posted 2019-02-11 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Venous Thromboses; Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism; Rheumatoid Arthritis; Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease; Psoriatic Arthritis
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism; Pulmonary Embolism; Arthritis, Rheumatoid; Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- People with inflammatory bowel disease: All individuals with an existing or incident diagnosis of IBD during the study period
  Interventions: Other: No intervention
- People with rheumatoid arthritis: All individuals with an existing or incident diagnosis of RA during the study period
  Interventions: Other: No intervention
- People with psoriatic arthritis: All individuals with an existing or incident diagnosis of IBD during the study period
  Interventions: Other: No intervention
- Controls: Age, gender and primary care practice matched individuals without an existing or incident diagnosis of IBD, RA, or PsA during the study period
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — A observation of outcomes in usual practice

SUMMARY:
Blood clots occurring in the legs and in the lungs are relatively common; they occur in around 3 in a 1000 people per year. They can cause disability and are also potentially life threatening. When a clot occurs in the legs it is called a deep vein thrombosis or DVT. When they occur in the lungs they are called a pulmonary embolism or PE. The risk for DVT and PE is higher in people with conditions which cause inflammation. The most common of these are inflammatory bowel disease (ulcerative colitis and Crohn's disease), rheumatoid arthritis, and psoriatic arthritis (a condition comprised of psoriasis and joint inflammation).

What is not known is how much higher the risk of DVT and PE is in these groups compared with people without inflammatory disease, and what causes the excess risk in these people. This study aims to assess the measure the exact increase in risk for DVT and PE in people with these inflammatory conditions and to identify which risk factors are most strongly associated with the increased risk. These data should help with an understand the causes of blood clot risk in these inflammatory conditions and in identify targets for reducing risk.

DETAILED DESCRIPTION:
Background

Venous thromboembolism (VTE), comprising pulmonary embolism (PE) and deep vein thrombosis (DVT), are common and associated with significant morbidity and mortality. VTE risk is higher in chronic inflammatory conditions including inflammatory bowel disease (IBD) and rheumatoid arthritis (RA) compared to the general population. Evidence for differential VTE risk in other inflammatory diseases, notably psoriatic arthritis (PsA) and vasculitis, is more limited. Risk factors for VTE have been described in the general population, but there has been little interrogation of VTE risk factors for individuals with chronic inflammatory conditions and their association with subsequent VTE.

Objective

This study aims to describe the prevalence of VTE risk and risk factors in individuals with systemic inflammatory disorders in a contemporary real-world population, by disease type (IBD, RA, and PsA) and relative to a control population without systemic inflammatory disease. In the same cohorts a further comparison will be performed of the influence of VTE risk factors on risk of VTE events in individuals with systemic inflammatory disorders.

Method

A retrospective cohort study will be performed to compare VTE risk and VTE risk factors in adults with IBD, RA, and PsA and matched controls between January 1, 1998 and January 1, 2018, within the Royal College of General Practitioners (RCGP) Research and Surveillance Centre (RSC) network. In the cohorts with and without inflammatory conditions estimate will be determined for the risk of VTE overall, and for PE and DVT separately, using unadjusted Cox proportional hazards models, stratified by matched set (exposed cohort versus unexposed cohort), to provide overall hazard ratios for the association with each outcome. Models will be subsequently adjusted for sociodemographic and clinical and VTE risk factors in multivariable analysis to explore potentially important associations with VTE. The same analyses for each autoimmune condition will be repeated separately. Prespecified sensitivity analyses will be performed to explore the robustness of any potential associations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥18) contributing to RCGP RCS primary care database between January 1, 1998 and January 1, 2018, will be eligible for inclusion

Exclusion Criteria:

* People with IBD which cannot be classified or is not ulcerative colitis or Crohn's disease will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The exposed cohort includes all individuals with an existing or incident diagnosis of IBD, RA or PsA (systemic inflammatory diseases) in the RCGP RSC over the study period. IBD, RA or PsA will be identified using Read diagnostic codes previously validated in UK primary care studies.
  The matched unexposed cohort will be defined by matching individuals in the exposed cohort with individuals never diagnosed with a systemic inflammatory disease either prior to or during the study period by age and sex. Unexposed individuals require at least 1 year of follow-up when matched to minimize the risk they had a non-recorded existing diagnosis of a systemic inflammatory disease of interest. Follow-up for each matched individual will begin at the start of follow-up of their matched counterpart.
Sampling Method: Non-Probability Sample
Enrollment: 266890 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McGovern, MD, Principal Investigator — Momentum Data
Locations (1):
- Momentum Data Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data is confidential but can be made available in an anonymised form to bone fide researchers subject to the required data protection training and other requirements. All data will remain behind a firewall and will only be available for access through a secured computer network.
Supporting Information: Study Protocol
Time Frame: The data will be available subject to approval for two years after the study publication date.
Access Criteria: Data sharing is subject to required data protection training and other requirements.

REFERENCES:
- [Derived] Irving PM, de Lusignan S, Tang D, Nijher M, Barrett K. Risk of common infections in people with inflammatory bowel disease in primary care: a population-based cohort study. BMJ Open Gastroenterol. 2021 Feb;8(1):e000573. doi: 10.1136/bmjgast-2020-000573. PMID 33597152
- [Derived] Galloway J, Barrett K, Irving P, Khavandi K, Nijher M, Nicholson R, de Lusignan S, Buch MH. Risk of venous thromboembolism in immune-mediated inflammatory diseases: a UK matched cohort study. RMD Open. 2020 Sep;6(3):e001392. doi: 10.1136/rmdopen-2020-001392. PMID 32994362

RESULTS

PARTICIPANT FLOW:
Groups:
- People With Ulcerative Colitis: All individuals with an existing or incident diagnosis of ulcerative colitis during the study period
  No intervention: A observation of outcomes in usual practice
- People With Crohn's Disease: All individuals with an existing or incident diagnosis of Crohn's during the study period
  No intervention: A observation of outcomes in usual practice
Period: Overall Study
Arm/Group | Controls | People With Ulcerative Colitis | People With Crohn's Disease | People With Psoriatic Arthritis | People With Rheumatoid Arthritis
Started | 213512 | 14182 | 9489 | 6297 | 23410
Completed | 213512 | 14182 | 9489 | 6297 | 23410
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- People With Crohn's Disease: All individuals with an existing or incident diagnosis of Crohn's disease during the study period
  No intervention: A observation of outcomes in usual practice
- Total: Total of all reporting groups
Arm/Group | Controls | People With Ulcerative Colitis | People With Crohn's Disease | People With Psoriatic Arthritis | People With Rheumatoid Arthritis | Total
Number analyzed (Participants) | 213512 | 14182 | 9489 | 6297 | 23410 | 266890
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years at study entry
  years | 51.7 (17.8) | 47.2 (17.0) | 41.8 (16.6) | 49.2 (13.8) | 59.0 (15.5) | 49.8 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128129 | 7056 | 5193 | 3204 | 16634 | 160216
  Male | 85383 | 7126 | 4296 | 3093 | 6776 | 106674
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9569 | 724 | 347 | 249 | 1114 | 12003
  Black | 4121 | 127 | 91 | 22 | 403 | 4764
  Mixed | 1483 | 85 | 67 | 44 | 150 | 1829
  Other | 1448 | 93 | 54 | 26 | 123 | 1744
  White | 148832 | 10099 | 6763 | 4727 | 17119 | 187540
  Missing | 48059 | 3054 | 2167 | 1229 | 4501 | 59010
Body mass index [Count of Participants; unit: Participants] — Body Mass Index (BMI) reported in kg/m2
  Participants
    Underweight (BMI ≤18.5) | 4704 | 368 | 536 | 60 | 607 | 6275
    Normal weight (BMI 18.5-25) | 73675 | 5721 | 4225 | 1576 | 7758 | 92955
    Overweight (BMI 25-30) | 67076 | 4352 | 2446 | 2131 | 7735 | 83740
    Obese (BMI ≥30) | 44303 | 2367 | 1386 | 2071 | 5787 | 55914
    BMI not recorded | 23754 | 1374 | 896 | 459 | 1523 | 28006
Smoking status [Count of Participants; unit: Participants]
  Non-Smoker | 94985 | 6328 | 3917 | 2522 | 8853 | 116605
  Current Smoker | 52035 | 2574 | 2914 | 1519 | 6063 | 65105
  Ex-Smoker | 63798 | 5147 | 2551 | 2232 | 8385 | 82113
  Smoking status not recorded | 2694 | 133 | 107 | 24 | 109 | 3067
Alcohol intake [Count of Participants; unit: Participants]
  Non-drinker | 36623 | 2371 | 1798 | 1035 | 5404 | 47231
  Within limits | 117939 | 7727 | 4917 | 3508 | 13164 | 147255
  Over recommended limits | 30096 | 2083 | 1228 | 1067 | 2767 | 37241
  Alcoholism | 3438 | 217 | 138 | 128 | 340 | 4261
  Alcohol level not recorded | 25416 | 1784 | 1408 | 559 | 1735 | 30902
Index of multiple deprivation (IMD) quintile [Count of Participants; unit: Participants] — Index of Multiple Deprivation (IMD) is a UK national deprivation measure of deprivation which is based on the patient postcode. IMD has been stratified into quintiles with IMD 1 representing most deprived and IMD 5 being the least deprived.
  Participants
    1 (most deprived) | 29144 | 1689 | 1324 | 803 | 3477 | 36437
    2 | 32323 | 2109 | 1518 | 919 | 3728 | 40597
    3 | 41379 | 2680 | 1901 | 1250 | 4739 | 51949
    4 | 50087 | 3475 | 2186 | 1452 | 5326 | 62526
    5 (least deprived) | 56209 | 3963 | 2350 | 1720 | 5651 | 69893
    IMD not recorded | 4370 | 266 | 210 | 153 | 489 | 5488

OUTCOME MEASURES:

1. Primary Outcome: Risk of Venous Thromboembolism (VTE)
Description: Number of participants with systemic inflammatory disorders developing VTE (a composite of pulmonary embolism (PE) and deep vein thrombosis (DVT)) compared to population controls.
Time Frame: A 20 year analysis period (1999-2018 inclusive)
Measure: Count of Participants; unit: Participants
Groups:
- People With Ulcerative Colitis (UC): All individuals with an existing or incident diagnosis of UC during the study period
  No intervention: A observation of outcomes in usual practice
- People With Crohn's Disease: All individuals with an existing or incident diagnosis of Crohn's disease during hte study period
Arm/Group | People With Ulcerative Colitis (UC) | People With Rheumatoid Arthritis | People With Psoriatic Arthritis | Controls | People With Crohn's Disease
Number analyzed (Participants) | 14182 | 23410 | 6297 | 213512 | 9489
Participants | 335 | 845 | 132 | 3804 | 220

2. Secondary Outcome: Risk of Pulmonary Embolism (PE)
Description: Number of participants with systemic inflammatory disorders developing PE compared to population controls.
Time Frame: A 20 year analysis period (1999-2018 inclusive)
Measure: Count of Participants; unit: Participants
Groups:
- People With Rheumatoid Arthritis (RA): All individuals with an existing or incident diagnosis of RA during the study period
  No intervention: A observation of outcomes in usual practice
- People With Psoriatic Arthritis (PsA): All individuals with an existing or incident diagnosis of PsA during the study period
  No intervention: A observation of outcomes in usual practice
- People With Crohn's Disease (CD): All individuals with an existing or incident diagnosis of CD during the study period
Arm/Group | People With Ulcerative Colitis (UC) | People With Rheumatoid Arthritis (RA) | People With Psoriatic Arthritis (PsA) | Controls | People With Crohn's Disease (CD)
Number analyzed (Participants) | 14182 | 23408 | 6297 | 213509 | 9489
Participants | 149 | 373 | 52 | 1737 | 98

3. Secondary Outcome: Risk of Deep Vein Thrombosis (DVT)
Description: Number of participants with systemic inflammatory disorders developing DVT compared to population controls.
Time Frame: A 20 year analysis period (1999-2018 inclusive)
Measure: Count of Participants; unit: Participants
Arm/Group | People With Ulcerative Colitis (UC) | People With Rheumatoid Arthritis (RA) | People With Psoriatic Arthritis (PsA) | Controls | People With Crohn's Disease (CD)
Number analyzed (Participants) | 14182 | 23408 | 6297 | 213510 | 9489
Participants | 207 | 542 | 89 | 2335 | 140

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study.
Arm/Group | Controls | People With Ulcerative Colitis | People With Crohn's Disease | People With Psoriatic Arthritis | People With Rheumatoid Arthritis
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT03835780/Prot_SAP_000.pdf